CLINICAL TRIAL: NCT07078084
Title: Laterality Training and Pain Drawings: A Randomized Controlled Trial
Brief Title: Laterality Training and Pain Drawings
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawaii Pacific University (Other)
Collaborators: Therapeutic Neuroscience Research Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5604202539
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Musculoskeletal Pain; Chronic Shoulder Pain; Chronic Knee Pain
Keywords: Chronic musculoskeletal pain; Shoulder pain; Knee pain; Laterality training; Left/right discrimination; Graded motor imagery; Pain neuroscience; Pain drawings
MeSH Terms: conditions — Shoulder Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model in which participants are randomly assigned to one of two groups: an intervention group receiving laterality training or a control group completing a non-therapeutic cognitive task. Each participant completes only one condition (no crossover), and pre- and post-intervention outcomes are compared between groups. This design allows researchers to evaluate the specific effects of laterality training on pain and pain-related body mapping.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laterality Training Intervention (Experimental): Participants in this arm will complete laterality training using the Recognise™ application. This involves identifying left or right hand or foot images (depending on the participant's pain location) displayed on a tablet. Each participant will complete 5 rounds of 60-second training with 60-second rest intervals between rounds. The activity is designed to engage cortical body maps and promote neuroplastic changes associated with reduced pain perception.
  Interventions: Behavioral: Laterality Training
- Sham Cognitive Task Comparator (Sham Comparator): Participants in this arm will complete a non-therapeutic cognitive activity by working independently on a standard word-based crossword puzzle for 10 minutes. This task is designed to match the duration and engagement level of the laterality training without influencing sensorimotor processing or cortical body maps. It serves as a sham comparator to help isolate the specific effects of the laterality training intervention
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Behavioral: Laterality Training — Participants complete a structured laterality training session using a tablet-based application that presents images of hands or feet. Depending on their pain location (shoulder or knee), participants identify whether each image shows a left or right body part. The session consists of 5 one-minute training bouts with 60-second rest intervals between each. The task is designed to engage and retrain cortical body maps associated with the painful region, based on principles of graded motor imagery. Participants are instructed to prioritize accuracy over speed.
  Other Names: Left/Right Discrimination Task
  Arms: Laterality Training Intervention
Other: Sham (No Treatment) — Participants in this arm will complete a non-therapeutic cognitive activity by working independently on a standard word-based crossword puzzle for 10 minutes. This task is designed to match the duration and engagement level of the laterality training without influencing sensorimotor processing or cortical body maps. It serves as a sham comparator to help isolate the specific effects of the laterality training intervention.
  Arms: Sham Cognitive Task Comparator

SUMMARY:
The goal of this clinical trial is to learn if laterality training (a type of brain-based therapy) can help reduce pain and change how people with chronic musculoskeletal pain experience and describe their pain. The study will focus on adults with shoulder or knee pain lasting longer than 6 months.

The main questions it aims to answer are:

Does laterality training lead to a reduction in self-reported pain levels?

Does laterality training reduce the area of the body that participants indicate as painful in their pain drawings?

Does laterality training improve accuracy and speed in left/right judgment tasks?

Researchers will compare participants who complete laterality training to those who complete a non-therapeutic cognitive task (a word puzzle) to see if laterality training changes pain drawings and improves pain outcomes.

Participants will:

Complete a pre-intervention assessment including pain ratings, pain drawings, and a left/right judgment test

Be randomly assigned to one of two groups:

Intervention group: Complete 5 one-minute sessions of laterality training using a tablet-based app called Recognise™, identifying left or right hand/foot images depending on the location of their pain

Control group: Complete a 10-minute crossword puzzle activity (non-therapeutic)

Complete the same assessments after the activity (pain ratings, pain drawings, left/right judgment test)

The study will take place at two outpatient physical therapy clinics. Participation involves a single session lasting approximately 30-45 minutes. There is no cost to participate, and no compensation is provided. Participation is voluntary, and all personal data will be kept confidential.

This research will help determine whether laterality training, a non-invasive brain-based technique, can reduce pain and improve quality of life in people with long-standing musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of chronic shoulder or knee pain lasting more than 6 months
* Able to read and understand English
* Willing to provide written informed consent

Exclusion Criteria:

* Visual impairments that would interfere with laterality training (e.g., blindness or significant difficulty with vision)
* Previous participation in laterality (left/right discrimination) training
* Unwilling or unable to participate in the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Drawing Area | Baseline and post-intervention (approximately 15 minutes after Baseline)
  Measured using a standardized body chart with a grid overlay. Participants mark areas of perceived pain, and the total number of grid squares marked is quantified to assess changes in spatial pain representation.

SECONDARY OUTCOMES:
Change in Left/Right Judgment Accuracy and Reaction Time | Baseline and post-intervention (approximately 15 minutes after Baseline)
  Assessed using the Recognise™ app. Participants complete two 60-second tests identifying left/right images of hands (shoulder pain) or feet (knee pain). Accuracy (%) and average response time (seconds per image) are recorded.
Change in Numeric Pain Rating Scale (NPRS) | Baseline and post-intervention (approximately 15 minutes after Baseline)
  Self-reported pain intensity measured using an 11-point numeric scale (0 = no pain, 10 = worst imaginable pain). This outcome assesses the immediate change in pain before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan P Louw, PhD, Principal Investigator — Therapeutic Neuroscience Research Group
Locations (2):
- United States (2):
  - Rock Valley Physical Therapy, Moline, Illinois
  - Rock Valley Physical Therapy, Davenport, Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanders NW, Mann NH 3rd, Spengler DM. Pain drawing scoring is not improved by inclusion of patient-reported pain sensation. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2735-41; discussion 2742-3. doi: 10.1097/01.brs.0000244674.99258.f9. PMID 17077744
- [Background] Matthews M, Rathleff MS, Vicenzino B, Boudreau SA. Capturing patient-reported area of knee pain: a concurrent validity study using digital technology in patients with patellofemoral pain. PeerJ. 2018 Mar 8;6:e4406. doi: 10.7717/peerj.4406. eCollection 2018. PMID 29568700
- [Background] Louw A, Farrell K, Zimney K, et al. Pain and Decreased Range of Motion in Knees and Shoulders: A Brief Sensory Remapping Intervention. Pain and Rehabilitation. 2017;Summer(43):20-30.
- [Background] Bowering KJ, O'Connell NE, Tabor A, Catley MJ, Leake HB, Moseley GL, Stanton TR. The effects of graded motor imagery and its components on chronic pain: a systematic review and meta-analysis. J Pain. 2013 Jan;14(1):3-13. doi: 10.1016/j.jpain.2012.09.007. Epub 2012 Nov 15. PMID 23158879
- [Background] Gurudut P, Godse AN. Effectiveness of graded motor imagery in subjects with frozen shoulder: a pilot randomized controlled trial. Korean J Pain. 2022 Apr 1;35(2):152-159. doi: 10.3344/kjp.2022.35.2.152. PMID 35354678